CLINICAL TRIAL: NCT01544270
Title: The Effects of Dietary Factors on Physiological Subjective Stress Responses in Cronically Stressed Subjects: a Randomised Clinical Trial
Brief Title: The Effects of Dietary Factors on Physiological Subjective Stress Responses
Acronym: AivoPro2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: SalWe Ltd. (Industry)
Responsible Party: Principal Investigator, Katri Peuhkuri, Principal investigator, postdoctoral reseacher, authorized nutritionist, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UH-SHOK-002
Record Dates: First submitted 2012-02-16; First posted 2012-03-05 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Stress
Keywords: milk protein; probiotics; stress; cortisol; heart beat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study product containing milk proteins (Active Comparator): Yoghurt-like milk-based product
  Interventions: Dietary Supplement: Yogurt-like snacks
- Study product containing probiotics (Active Comparator): Yoghurt-like milk-based product
  Interventions: Dietary Supplement: Yogurt-like snacks
- Control product (Placebo Comparator): Yoghurt-like milk-based product without supplemented nutrients
  Interventions: Dietary Supplement: Yogurt-like snacks

INTERVENTIONS:
Dietary Supplement: Yogurt-like snacks — twice a day 120 g for four weeks

SUMMARY:
The study aims to investigate the role of dietary factors in chronically stressed subjects. Previous studies have shown that milk proteins, B vitamins and probiotics may influence on subjective well-being in stressed subjects.

ELIGIBILITY:
Inclusion Criteria:

* STAI points 40-65
* BMI 18-30 kg/m2
* healthy

Exclusion Criteria:

* Gastrointestinal disease, diabetes or any other significant major medical morbidity
* milk allergy
* smoking
* excess use of alcohol
* pregnancy and breast feeding
* waist circumference males >102 cm, females >88 cm
* no medication or dietary supplements influencing measured responses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Subjective well-being | baseline and 4 weeks
  Change in stress and mood states measured by State-trait anxiety inventory (STAI) and modified Profile of Mood States (POMS) at baseline and after 4 wk intervention

SECONDARY OUTCOMES:
Physiological measurements | baseline and 4 weeks
  Change in salivary cortisol, blood pressure, heart beat variability, sleep and inflammatory markers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Institute of Biomedicine, Helsinki, Finland

REFERENCES:
- [Derived] Jaatinen N, Korpela R, Poussa T, Turpeinen A, Mustonen S, Merilahti J, Peuhkuri K. Effects of daily intake of yoghurt enriched with bioactive components on chronic stress responses: a double-blinded randomized controlled trial. Int J Food Sci Nutr. 2014 Jun;65(4):507-14. doi: 10.3109/09637486.2014.880669. Epub 2014 Feb 4. PMID 24490888